CLINICAL TRIAL: NCT05048602
Title: Drug-induced Brugada Syndrome Research Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Vincenzo Russo, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 07082021
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Brugada Syndrome; Arrhythmia; ICD
MeSH Terms: conditions — Brugada Syndrome; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All patients with drug-induced Brugada syndrome who are evaluated and followed at each participating centers will be recorded in this register. Within this register a characterization of patients and therapy will be done. Prognostic factors of adefined clinical relevant endpoints will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with drug-induced Brugada Syndrome

Exclusion Criteria:

* Missing Informed Consent Form
* Missing Contact Informations for Follow up

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with drug-induced Brudaga Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-09-07 (Estimated); Study Completion 2025-09-07 (Estimated)

PRIMARY OUTCOMES:
Sudden Cardiac Death | 1 year
  Unexpected death due to cardiac causes that occurs in a short time period.
Appropriate ICD Therapies | 1 year
  Antitachycardia pacing therapy or shock delivered by ICD for device detected ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Russo, MD PhD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- Vincenzo Russo, Naples, Napoli, Italy